CLINICAL TRIAL: NCT06225999
Title: A Single-arm Multicentre Phase 2 Study of Irinotecan Liposome Injection, Oxaliplatin, 5-fluorouracil/Levoleucovorin in Japanese Participants Who Have Not Previously Received Therapy for Metastatic Adenocarcinoma of the Pancreas
Brief Title: Phase 2 Study of Irinotecan Liposome Injection, Oxaliplatin, 5-fluorouracil/Levoleucovorin in Japanese Participants Not Previously Treated for Metastatic Adenocarcinoma of the Pancreas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S095013-169
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Adenocarcinoma of the Pancreas
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposome Injection in combination with oxaliplatin, 5-FU and LLV (Experimental)
  Interventions: Drug: Irinotecan liposome injection (S095013); Drug: Oxaliplatin; Drug: LLV (levoisomer form of leucovorin); Drug: 5- FU (5-Fluorouracil)

INTERVENTIONS:
Drug: Irinotecan liposome injection (S095013) — Irinotecan liposome injection (S095013) will be administered via intravenous (IV) infusion on days 1 and 15 of each 28-day cycle.
  Other Names: MM-398; Nal-IRI; BAX2398; PEP02; liposomal irinotecan
Drug: Oxaliplatin — Oxaliplatin will be administered via intravenous (IV) infusion on days 1 and 15 of each 28-day cycle.
Drug: LLV (levoisomer form of leucovorin) — LLV will be administered via intravenous (IV) infusion on days 1 and 15 of each 28-day cycle.
Drug: 5- FU (5-Fluorouracil) — 5-FU will be administered via intravenous (IV) infusion on days 1 and 15 of each 28-day cycle.

SUMMARY:
This study is to assess the anti-tumour activity, safety and tolerability of irinotecan liposome injection (S095013) in combination with oxaliplatin, 5-Fluorouracil (5-FU) and levoisomer form of leucovorin (LLV). S095013, oxaliplatin, 5-FU and LLV will be administered on days 1 and 15 of each 28-day cycle. Cycles will continue until clinical or radiological progressive disease, unacceptable study medication-related toxicity or withdrawal from study. During the treatment period participants will have study visits on day 1, 3, 15, and 17 of each cycle, some of which may occur as a home visit. At least 30 days after treatment has ended a end of treatment visit will occur and then participants will be followed for survival every month via telephone or email until death or end of the study. Study visits may include questionnaires, blood and urine tests, ECG, vital signs, physical examination, and administration of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating female ≥ 18 years of age.
* Histologically or cytologically confirmed adenocarcinoma of the pancreas that has not been previously treated in the metastatic setting.
* Initial diagnosis of metastatic disease (as per American Joint Committee on Cancer 8th Edition [AJCC 2017]) must have occurred ≤ 6 weeks prior to screening.
* Participant has one or more metastatic lesions measurable by CT-scan (or MRI), if the participant is allergic to CT contrast media, according to RECIST Version 1.1 criteria.
* ECOG PS of 0 or 1 at screening and within 7 days prior to first dosing.
* Participant has adequate hematological, biochemical, hepatic, and renal function parameters.

Exclusion Criteria:

* Prior treatment of pancreatic cancer in the metastatic setting with surgery, radiotherapy, chemotherapy or investigational therapy (palliative surgery, palliative radiotherapy and placement of biliary stent/tube are permitted).
* Prior treatment of pancreatic adenocarcinoma with chemotherapy in the adjuvant setting, except those where at least 12 months have elapsed since completion of the last dose and no persistent treatment-related relevant toxicities are present.
* Participant has only locally advanced disease.
* Known hypersensitivity to any of the components of irinotecan liposome injection, other liposomal products, or any components of 5-FU, LLV or oxaliplatin products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response (OR) | Through the end of study treatment (approximately 16 months after study start)
  OR is defined as complete response (CR) or partial response (PR), as assessed by the independent central review (ICR) per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Locations (14):
- Japan (14):
  - National Cancer Center Hospital East (003), Kashiwa, Chiba
  - Chiba University Hospital (015), Chiba
  - Chiba Cancer Center (011), Chiba
  - National Hospital Organization Shikoku Cancer Center (013), Ehime
  - National Hospital Organization Kyushu Cancer Center (005), Fukuoka
  - Kanazawa University Hospital (008), Ishikawa
  - Kanagawa Cancer Center (002), Kanagawa
  - Aichi Cancer Center (007), Nagoya
  - Osaka International Cancer Institute (009), Osaka
  - Saitama Cancer Center (012), Saitama
  - Hokkaido University Hospital (004), Sapporo
  - National Cancer Center Hospital (001), Tokyo
  - The Cancer Institute Hospital of JFCR (006), Tokyo
  - Yamaguchi University Hospital (010), Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/

REFERENCES:
- [Derived] Ikeda M, Okusaka T, Ueno M, Ozaka M, Satoi S, Skanji D, Martin-Fernandez L, Amellal N, Furuse J. NALIRIFOX in Japanese treatment-naive patients with metastatic pancreatic adenocarcinoma: an open-label, phase II trial design. Future Oncol. 2025 Apr;21(8):959-965. doi: 10.1080/14796694.2025.2469467. Epub 2025 Feb 22. PMID 39987459